CLINICAL TRIAL: NCT04080674
Title: Studying the Role of the Basal Ganglia in Motor Symptoms Using Deep Brain Stimulation
Brief Title: Using DBS to Probe Basal Ganglia Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 271953
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Parkinson's Disease; Tremor; Dystonia
MeSH Terms: conditions — Parkinson Disease; Tremor; Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's disease: 30 participants
  Interventions: Other: Feed-back controlled deep brain stimulation
- Essential Tremor: 10 participants
  Interventions: Other: Feed-back controlled deep brain stimulation
- Dystonia: 20 participants
  Interventions: Other: Feed-back controlled deep brain stimulation

INTERVENTIONS:
Other: Feed-back controlled deep brain stimulation — Feed-back controlled deep brain stimulation

SUMMARY:
This study will probe the function of collections of neurons deep in the brain termed the basal ganglia It will investigate the role of the basal ganglia in how and why movement is disrupted in conditions like Parkinson's disease, Dystonia and Essential Tremor. Deep brain recording and stimulation will be used to probe the basal ganglia's contribution. Patients with relatively severe movement disorders may have electrodes implanted in the basal ganglia so that stimulation can be delivered chronically as a form of therapy. Studying these patients allows researchers (a) to record brain activity from these electrodes in the basal ganglia during symptoms related to abnormal motor control and (b) to stimulate the same electrodes while patients experience symptoms. Like this they can see what aspects of the activity of groups of nerve cells in the basal ganglia are associated with which symptoms and also establish that these aspects of activity help cause linked symptoms. This means studying patients just after electrode implantation, while the leads from the electrodes may still be available for hooking up to external recording and stimulating devices. Understanding how the activity of groups of nerve cells in the basal ganglia controls movement may help us develop improved treatments.

DETAILED DESCRIPTION:
This study investigates how the basal ganglia contribute to motor symptoms like tremor, bradykinesia and muscle spasm. The basic research approach is to record from sites in the basal ganglia whilst patients are symptomatic, so that brain waves can be correlated with symptoms/signs. Once a brain wave is implicated in an aspect of abnormal movement, the researchers can try and confirm its central role in function or dysfunction by triggering stimulation whenever the brain wave is picked up. For stimulation the researchers will use the same high frequency stimulation (130 Hz) as used clinically, as this is thought to effectively suppress neural activity at the stimulation site. Thus, if a given brain wave is important in, for example, slowing movement, then by triggering stimulation whenever this brain wave is big it can be expected that movement speed will be increased.

The investigators hope to follow this two-stage procedure to document the role of the different brain activities picked up from basal ganglia sites in driving tremor, muscle spasm and slowness of movement in patients with Parkinson's disease, dystonia and essential tremor. This study is important, as if the researchers can alter brain function and specific symptoms with stimulation they can use the same form of feedback-controlled stimulation as a potentially efficient form of treatment. Conventional deep brain stimulation delivers fixed stimulation all of the time. For example, researchers are beginning to see that stimulation control based on feedback from beta activity in the basal ganglia may have advantages over conventional continuous deep brain stimulation in treating Parkinson's disease.

The current study is particularly interested in the processes contributing to slowness (bradykinesia) and rigidity (stiffness) in patients with Parkinson's disease, tremor in patients with Parkinson's disease and Essential Tremor, and muscle spasms in patients with dystonia.

1. Bradykinesia and Rigidity in patients with Parkinson's disease Here there is already evidence that these impairments are associated with beta frequency band activity (~20Hz). Such activity is exaggerated in patients with Parkinson's disease in whom it comes in bursts lasting several hundred milliseconds or even longer. The investigators have already shown that by triggering stimulation when bursts of beta activity occur they can speed up movement and reduce rigidity. In the present study they are interested in (a) determining whether it is necessary to trigger off beta bursts or whether it is sufficient to trigger off the general level of beta activity (ie averaged over long periods), (b) whether if it is necessary to trigger off all beta bursts, or is it just the long bursts that need to be triggered off, and (c) whether triggered stimulation is also sufficient to control tremor where this is a co-existent symptom. Exploration of these issues requires the investigators to record basal ganglia activity (the feedback) and to deliver stimulation, whilst varying how the feedback is processed before driving the stimulation. In engineering terms the investigators vary the signal processing and control policy details, but the net result is feedback-controlled deep brain stimulation. Note that the investigators only control the amplitude of stimulation within a clinically determined range that goes no higher than the threshold for eliciting side-effects. All the remaining stimulation parameters, e.g. frequency and pulse width, are set to standard clinical settings.
2. Tremor in patients with Parkinson's disease or Essential Tremor Here the evidence that tremor is associated with a discrete brain activity is less robust, although oscillations at tremor frequency (and twice this) are suspected of playing a role. In conditions where the investigators are unsure of the exact nature of the factors contributing to a state, in this case tremor, they often use machine learning to find the relevant factors. Here the investigators propose to record both basal ganglia activity and tremor in the limbs and then use these with machine learning algorithms to point out the relevant combination of signals associated with tremor. The investigators can then use machine learning outputs to tell them how to control tremor with stimulation, whilst interrogating the weights of the inputs to the machine learning algorithms to deduce the important relationships. As above, they will explore the optimal signal processing and control policy details, but the net result is feedback-controlled deep brain stimulation. Note that they only control the amplitude of stimulation within a clinically determined range that goes no higher than the threshold for eliciting side-effects. All the remaining stimulation parameters, e.g. frequency and pulse width, are set to standard clinical settings.
3. Involuntary muscle spasms in patients with Dystonia Here the evidence that muscle spasms are associated with a discrete brain activity is also relatively weak, although oscillations at theta-alpha frequencies (5-12 Hz) are suspected of playing a role. The investigators propose to record both basal ganglia activity and muscle spasms in the body and then use these with machine learning algorithms to point out the relevant combination of signals associated with muscle spasms. They can then use machine learning outputs to tell them how to control muscle spasms with stimulation. As above, the investigators will explore the optimal signal processing and control policy details, but the net result is feedback-controlled deep brain stimulation. Note that they only control the amplitude of stimulation within a clinically determined range that goes no higher than the threshold for eliciting side-effects. All the remaining stimulation parameters, e.g. frequency and pulse width, are set to standard clinical settings.

Techniques to be used

Our study involves several techniques:

1. Evaluation of symptoms using standard clinical rating scales e.g Part III motor UPDRS, Unified dyskinesia rating scale and speech intelligibility test in patients with Parkinson's disease; essential tremor rating assessment scale (TETRAS) for patients with essential tremor; Burke Fahn Marsden dystonia rating scale (BFMDRS) for patients with dystonia. The performance of these rating scales will also be videoed for off-line review.
2. Recording of peripheral symptoms like movement speed, tremor or spasm with standard techniques e.g. recording joystick movement speed, recording tremor and other movements with the bradykinesia akinesia incoordination test, skin mounted accelerometers and skin mounted electromyographic (EMG) electrodes. These are standard, non-invasive techniques that do not involve any side-effects of discomfort.
3. Recording of EEG using scalp mounted electrodes. This is a standard, non-invasive technique that does not involve any side-effects or discomfort. However, there is an important caveat here that as these patients will have recent surgical scars on their scalps these will avoided so that no electrode is applied to the scalp within 4 cm of any wound. EEG electrodes are applied to the scalp with a conductive paste which helps hold them in place. Sometimes, where lack of hair allows, the investigators bolster that attachment with some tape. There is no increase in infection risk due to recordings in patients with externalised deep brain stimulation leads.
4. Recordings of depth EEG from the deep brain stimulation electrodes implanted in to the brain by the surgeon for standard clinical therapy. As these are passive recordings there are no side-effects or risks. Recordings in 2-4 will be performed using an amplifier that holds a certification mark that indicates conformity with health, safety, and environmental protection standards for products sold within the European Economic Area.
5. Stimulation of the deep brain stimulation electrodes implanted in to the brain by the surgeon for standard clinical therapy. Stimulation can cause side-effects, so importantly the investigators will only deliver stimulation in the form and range used clinically, taking care to always remain below the threshold for side-effects. Stimulation will be delivered through an in-house, custom-built, battery-supplied, bilateral stimulator that does not hold a certification mark that indicates conformity with health, safety, and environmental protection standards for products sold within the European Economic Area. Nevertheless, it has been fully safety tested. The stimulator is an updated version of that used for several past studies that have been reviewed and approved by the United Kingdom National Research Ethics Service Committee South Central. To allow for stimulation return, the amplifier is connected to a conducting pad placed over the neck. Periodic impedance checks will ensure this connection is robust through the course of the experiment.

Participants will be given the choice to undergo the study without their usual medication for their motor symptoms or with such medication. The former state is preferred to facilitate the demonstration of a link between neural activities and symptoms, but the final decision will be down to the participant. Symptoms may be worse with the temporary withdrawal of medication, but most participants will be familiar with this as a result of forgetting their medication in the past or because their medication was temporarily withdrawn as part of a clinical test like the levodopa challenge.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 to 80 years old.
* Diagnosed with Parkinson's disease, Essential Tremor or Dystonia.
* Undergoing two-stage surgery for deep brain stimulation as therapy for their movement disorder.

Exclusion Criteria:

* Cognitive impairment (judged by the clinician on the care team or in the research team as a participant not having sufficient mental capacity to understand the study and its requirements). This includes anyone who, in the opinion of clinicians on the care team or clinicians in the research team, is unlikely to retain sufficient mental capacity for the duration of their involvement in the study.
* Intracranial bleeding, confusion, cerebrospinal fluid leak or any other complication after the first stage of surgery.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing staged implantation of DBS electrodes
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Kinematic recordings | During stimulation
  Change in kinematic data
Electromyographic signals | During stimulation
  Change in electromyographic data
Disease relevant rating scale | During stimulation
  Change in disease relevant rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brown, MD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Undecided